CLINICAL TRIAL: NCT04790526
Title: Dose Response of Eccentric Exercises on Glycemic Control in Type ii Diabetes Mellitus
Brief Title: Dose Response of Eccentric Exercise on Glycemic Control in Type II Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RiphahIU M Faheem Afzal
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Type II Diabetes Mellitus
Keywords: Dose response; Eccentric exercise; Type II Diabetes Mellitus; Glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): This group includes 15 male participants who will be given 10 minutes of warm and cool down sessions that includes stationary bicycle without resistance and stretching. Intervention will be given with declination of treadmills at 16 degree and 3 session of 10 minutes duration will be given with 1 minutes of rest in each group. Intervention will be given for 3 sessions per week up to 12 weeks.
  Interventions: Other: Eccentric Exercises Dose
- Group B (Experimental): This group includes 15 female participants who will be given 10 minutes of warm and cool down sessions that includes stationary bicycle without resistance and stretching. Intervention will be given with declination of treadmills at 16 degree and 3 session of 10 minutes duration will be given with 1 minutes of rest in each group. Intervention will be given for 3 sessions per week up to 12 weeks.
  Interventions: Other: Eccentric Exercises Dose
- Group C (Experimental): This group includes 15 male participants who will be given 10 minutes of warm and cool down sessions that includes stationary bicycle without resistance and stretching. Intervention will be given with declination of treadmills at 16 degree and 3 session of 10 minutes duration will be given with 1 minutes of rest in each group. Intervention will be given for 5 sessions per week up to 12 weeks.
  Interventions: Other: Eccentric Exercises Dose
- Group D (Experimental): This group includes 15 female participants who will be given 10 minutes of warm and cool down sessions that includes stationary bicycle without resistance and stretching. Intervention will be given with declination of treadmills at 16 degree and 3 session of 10 minutes duration will be given with 1 minutes of rest in each group. Intervention will be given for 5 sessions per week up to 12 weeks.
  Interventions: Other: Eccentric Exercises Dose

INTERVENTIONS:
Other: Eccentric Exercises Dose — Eccentric exercise will be done treadmill in control environment. The treadmill will be declined to 16 degree and 3 sessions of 10 minutes duration will be given wit 1 minute of rest in each session. 10 minutes of warm up and cool down session will be given that includes stretching and stationary bicycle with out any resistance

SUMMARY:
The major aim of this project to check the dose response of eccentric exercise in reduction of glycemic index in type II Diabetes Mellitus. This study aim to check the effect of eccentric exercises on Glycemic index, quality of life, strength, exertion, balance and proprioception in type II Diabetes Mellitus patients

DETAILED DESCRIPTION:
From the last three decades, the diabetes mellitus progress quadrupled.The International Diabetes Federation (IDF) approximate that 1 in 11 adults with age between 20 to 79 years have diabetes mellitus. Almost 90 percent of patients diagnosed with Diabetes Mellitus are type 2 diabetes mellitus patients. According to the World Health Organization, Diabetes mellitus could be 7th leading cause of death. Type II Diabetes Mellitus (T2DM) increase progressively that affect around 25 million people in Europe and major public health issue for middle income countries. It is proposed that the prevalence of diabetes mellitus will increase up to 67% in middle-income countries from 2010 to 2030. In Pakistan, the Type II Diabetes Mellitus prevalence in 2018 is 11.77%. The prevalence is more in male as compared to females and urban area have 14.81 percent as compared to rural area.

The genetic architecture might partially determine an individual's response to environmental changes.The risk factors of Type II Diabetes Mellitus include obesity, ageing, behavioral and environment factors, diet and lifestyle. School-age children had also warned of a rise in childhood obesity in Pakistan, which is considered a strong risk factor in diabetic patients. The major cause of Type II Diabetes Mellitus is deficiency or loss of insulin. Brain utilize glucose as source of energy and when brain is unable to maintain integrity, Many physiological mechanism initiates to reduce and limit the effect of hypoglycemia.The response of human body in reaction to reduce glucose level causes lowering the secretion of insulin and release counter-regulatory hormone.Diabetes mellitus have strong correlation for reduction in muscular strength and functional status.

A recent study on global burden of diseases, Diabetes mellitus considered as ninth major cause of reduced life expectancy. A study conducted decades ago concluded that 3.96 million deaths occur due to diabetes mellitus with aged between 20-79 years. According to the International Diabetes Federation, the number and complications of diabetes mellitus increase rapidly up to 5.0 million deaths due to metabolic disorder.The prevalence of disability occurrence due to diabetes mellitus increase significantly since 3 decades ago. According to the global burden of Disease, Injuries and Risk factor statement, the 10th most common factor of disability was fasting level of glucose in 1990, 4th common cause till 2005 and 3rd common cause in 2015.45.8 percent of diabetes mellitus patients were approximately not diagnosed. Those patient who are not diagnosed have more risk of complication as compared to those who are diagnosed and start intervention. Medical expenditure of diabetes mellitus patients increases three times more than general population.The cases of people living suffering from Type II Diabetes Mellitus increase quadrupled between 1980 and 2014 globally. Adults who have diagnosed diabetes mellitus enhance to 20 percent from 2010 to 2030 and predicted to increase rapidly up to 69 percent. In Asia, the epidemic of Type II Diabetes Mellitus progress very rapidly and characterized by onset at a lower BMI and younger age than in Western populations. An average cost for the treatment of Diabetes Mellitus in Pakistan ranges from 650 to 20000 PKR.

ELIGIBILITY:
Inclusion Criteria:

Cleared by a general practitioner to attend the training program Sedentary patients with controlled type 2 diabetes, according to the definition of the American Diabetes Association.

Participants were untrained and had not engaged in resistance or aerobic exercise within 6 months prior to beginning the study.

Age between 45-65 Years. BMI should be 18.5-34.9 kg/m2.

Exclusion Criteria:

Participants with GIT disturbance (Gastroparesis and non-alcoholic fatty liver disease) will be excluded from the study.

Participants with any kind of Musculo-skeletal injury will be excluded from the study.

Participants with Stage II hypertension according to AHA guidelines. Participants who use tobacco products within the previous 6 months. Participants who take any type of systematic medication within the previous 6 months except diabetes.

Participants with any symptoms of neuropathy, retinopathy or nephropathy will be excluded

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with Type II Diabetes Mellitus
Enrollment: 59 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Glucometer | 12 week
  Glucometer will use to monitor glucose before and after the intervention. Glucometer have poor validity and reliability but consider medical tool for the management of diabetes.
HBA1c | 0 week and 12th week
  The A1C test is the most common diagnostic and screening tool used for Type II Diabetes Mellitus (T2DM) management and research

SECONDARY OUTCOMES:
WHO-QOL (BREF-Urdu version) | 0 week,4th week,8th week and 12th week
  WHOQOL-BREF is a short version of WHOQOL-100 developed under the supervision of World Health Organization.
Six Minutes' Walk Test | 0 week,4th week,8th week and 12th week
  The Six-minute walk test (6-MWT) is also a widely used method for evaluating cardiopulmonary performance
Dynamometer | 0 week,4th week,8th week and 12th week
  Commonly used devices that measure strength of body and include isometric lower limb muscle strength include dynamometers
Borg's Exertion Scale | 0 week,4th week,8th week and 12th week
  Borg scale of exertion is widely used in patients to identify intensity of exercise
BERG Balance Scale | 0 week,4th week,8th week and 12th week
  This scale is commonly used to check risk fall in elderly population
Joint error position test | 0 week,4th week,8th week and 12th week
  Joint position error (JPE) is widely used to quantitatively assess proprioception in rehabilitation and sport science

CONTACTS AND LOCATIONS:
Overall Officials: M Faheem Afzal, *PhD, Principal Investigator — Lahore Medical and Dental College
Locations (1):
- Rehabilitation Department, PSRD Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF DIABETES ATLAS [Internet]. 10th edition. Brussels: International Diabetes Federation; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK581934/ PMID 35914061
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in diabetes since 1980: a pooled analysis of 751 population-based studies with 4.4 million participants. Lancet. 2016 Apr 9;387(10027):1513-1530. doi: 10.1016/S0140-6736(16)00618-8. Epub 2016 Apr 6. PMID 27061677
- [Background] Holman N, Young B, Gadsby R. Current prevalence of Type 1 and Type 2 diabetes in adults and children in the UK. Diabet Med. 2015 Sep;32(9):1119-20. doi: 10.1111/dme.12791. No abstract available. PMID 25962518
- [Background] Bruno G, Runzo C, Cavallo-Perin P, Merletti F, Rivetti M, Pinach S, Novelli G, Trovati M, Cerutti F, Pagano G; Piedmont Study Group for Diabetes Epidemiology. Incidence of type 1 and type 2 diabetes in adults aged 30-49 years: the population-based registry in the province of Turin, Italy. Diabetes Care. 2005 Nov;28(11):2613-9. doi: 10.2337/diacare.28.11.2613. PMID 16249528
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] The Federal Ministry of Health and Women, Division IV (2006) European Union conference on prevention of type 2 diabetes, Vienna.
- [Background] Ogurtsova K, da Rocha Fernandes JD, Huang Y, Linnenkamp U, Guariguata L, Cho NH, Cavan D, Shaw JE, Makaroff LE. IDF Diabetes Atlas: Global estimates for the prevalence of diabetes for 2015 and 2040. Diabetes Res Clin Pract. 2017 Jun;128:40-50. doi: 10.1016/j.diabres.2017.03.024. Epub 2017 Mar 31. PMID 28437734
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Basit A, Fawwad A, Qureshi H, Shera AS; NDSP Members. Prevalence of diabetes, pre-diabetes and associated risk factors: second National Diabetes Survey of Pakistan (NDSP), 2016-2017. BMJ Open. 2018 Aug 5;8(8):e020961. doi: 10.1136/bmjopen-2017-020961. PMID 30082350
- [Background] Chatterjee S, Khunti K, Davies MJ. Type 2 diabetes. Lancet. 2017 Jun 3;389(10085):2239-2251. doi: 10.1016/S0140-6736(17)30058-2. Epub 2017 Feb 10. PMID 28190580
- [Background] O'Rahilly S. Human genetics illuminates the paths to metabolic disease. Nature. 2009 Nov 19;462(7271):307-14. doi: 10.1038/nature08532. PMID 19924209
- [Background] Sui X, Hooker SP, Lee IM, Church TS, Colabianchi N, Lee CD, Blair SN. A prospective study of cardiorespiratory fitness and risk of type 2 diabetes in women. Diabetes Care. 2008 Mar;31(3):550-5. doi: 10.2337/dc07-1870. Epub 2007 Dec 10. PMID 18070999
- [Background] Misra A, Vikram NK, Sharma R, Basit A. High prevalence of obesity and associated risk factors in urban children in India and Pakistan highlights immediate need to initiate primary prevention program for diabetes and coronary heart disease in schools. Diabetes Res Clin Pract. 2006 Jan;71(1):101-2. doi: 10.1016/j.diabres.2005.06.006. Epub 2005 Aug 19. No abstract available. PMID 16112243
- [Background] Chen L, Pei JH, Kuang J, Chen HM, Chen Z, Li ZW, Yang HZ. Effect of lifestyle intervention in patients with type 2 diabetes: a meta-analysis. Metabolism. 2015 Feb;64(2):338-47. doi: 10.1016/j.metabol.2014.10.018. Epub 2014 Oct 23. PMID 25467842
- [Background] Mitrakou A, Ryan C, Veneman T, Mokan M, Jenssen T, Kiss I, Durrant J, Cryer P, Gerich J. Hierarchy of glycemic thresholds for counterregulatory hormone secretion, symptoms, and cerebral dysfunction. Am J Physiol. 1991 Jan;260(1 Pt 1):E67-74. doi: 10.1152/ajpendo.1991.260.1.E67. PMID 1987794
- [Background] King P, Macdonald IA: Normal glucose metabolism and response to hypoglycaemia. In Hypoglycaemia in Clinical Diabetes. Frier BM, Fisher BM, Eds. Chichester, U.K., John Wiley and Sons, 1999, p. 29-54.
- [Background] Fanelli C, Pampanelli S, Epifano L, Rambotti AM, Di Vincenzo A, Modarelli F, Ciofetta M, Lepore M, Annibale B, Torlone E, et al. Long-term recovery from unawareness, deficient counterregulation and lack of cognitive dysfunction during hypoglycaemia, following institution of rational, intensive insulin therapy in IDDM. Diabetologia. 1994 Dec;37(12):1265-76. doi: 10.1007/BF00399801. PMID 7895957
- [Background] Nishitani M, Shimada K, Sunayama S, Masaki Y, Kume A, Fukao K, Sai E, Yamashita H, Ohmura H, Onishi T, Shioya M, Sato H, Shimada A, Yamamoto T, Amano A, Daida H. Impact of diabetes on muscle mass, muscle strength, and exercise tolerance in patients after coronary artery bypass grafting. J Cardiol. 2011 Sep;58(2):173-80. doi: 10.1016/j.jjcc.2011.05.001. Epub 2011 Jul 13. PMID 21741799
- [Background] Anton SD, Karabetian C, Naugle K, Buford TW. Obesity and diabetes as accelerators of functional decline: can lifestyle interventions maintain functional status in high risk older adults? Exp Gerontol. 2013 Sep;48(9):888-97. doi: 10.1016/j.exger.2013.06.007. Epub 2013 Jul 4. PMID 23832077
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Roglic G, Unwin N. Mortality attributable to diabetes: estimates for the year 2010. Diabetes Res Clin Pract. 2010 Jan;87(1):15-9. doi: 10.1016/j.diabres.2009.10.006. Epub 2009 Nov 14. PMID 19914728
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] GBD 2015 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 79 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1659-1724. doi: 10.1016/S0140-6736(16)31679-8. PMID 27733284
- [Background] Rubin RJ, Altman WM, Mendelson DN. Health care expenditures for people with diabetes mellitus, 1992. J Clin Endocrinol Metab. 1994 Apr;78(4):809A-809F. doi: 10.1210/jcem.78.4.8157701.
- [Background] Kong AP, Xu G, Brown N, So WY, Ma RC, Chan JC. Diabetes and its comorbidities--where East meets West. Nat Rev Endocrinol. 2013 Sep;9(9):537-47. doi: 10.1038/nrendo.2013.102. Epub 2013 May 28. PMID 23712250
- [Background] Hussain M, Naqvi SB, Khan MA, Rizvi M, Alam S, Abbas A, Akram MU. Direct cost of treatment of diabetes mellitus type 2 in Pakistan. Int J Pharm Pharm Sci. 2014;6(11):261-4.